CLINICAL TRIAL: NCT07237087
Title: Effects of Heat Application and Percussion Therapy on Masseter Muscle Stiffness Measured With Ultrasound Shear Wave Elastography
Brief Title: Masseter Muscle Stiffness After Heat Application and Percussion Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2025-00295
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
Keywords: TMD; shear wave elastography; ultrasound; elastography; Elasticity Imaging Techniques; heat pad; massage gun; heat treatment; percussion massage
MeSH Terms: conditions — Fever | interventions — Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: First massage gun, then heat treatment (Experimental): The massage gun is the new treatment (experimental). Heat treatment is already commonly used for muscle stiffness and could be considered an active comparator. However, since its specific effects on the masseter muscle are not well established, it may also be classified as experimental.
  Interventions: Device: massage gun; Device: heat treatment
- Group B: first heat treatment, then massage gun (Experimental): The massage gun is the new treatment (experimental). Heat treatment is already commonly used for muscle stiffness and could be considered an active comparator. However, since its specific effects on the masseter muscle are not well established, it may also be classified as experimental.
  Interventions: Device: massage gun; Device: heat treatment

INTERVENTIONS:
Device: massage gun — The massage gun used in this study will be equipped with a soft attachment designed for use on the face, ensuring safe and comfortable application to the masseter muscle.
Device: heat treatment — The heat treatment will be applied for 20min.
  Other Names: heat pad; heating pad

SUMMARY:
The purpose of this study is to evaluate the changes in the stiffness of the masseter muscle (a jaw muscle) before and after two types of treatment: applying commercial heat pads or using a commercial massage gun.

We will measure the muscle stiffness on the surface of the muscle using a special ultrasound probe, with a method called shear wave elastography.

When this muscle is too stiff, it's often linked to jaw pain and problems with the jaw joint - a condition known as Temporomandibular Disorder (TMD).

The goal is to find better treatment options for people with TMD and to collect data using this imaging technique.

DETAILED DESCRIPTION:
In our study, participants will be randomly assigned to one of two groups. This is important to ensure reliable results and is called randomization.

The two groups are as follows:

Group A:

First, the stiffness of the masseter muscle in the cheek is measured using ultrasound. Then, we will assess the mouth opening, the muscle's sensitivity to pressure, bite force, and chewing efficiency using several short tests. After that, the masseter muscle will be treated with a massage gun with a soft attachment for 2 minutes. All tests will be repeated after the treatment.

Group B:

First, the stiffness of the masseter muscle in the cheek is measured using ultrasound. Then, we will assess the mouth opening, the muscle's sensitivity to pressure, bite force, and chewing efficiency using several short tests. After that, the masseter muscle will be treated with a heat pad for 20 minutes. The heat pad will be held in place with a strap, and participants may sit and read or relax during the treatment. All tests will be repeated after the treatment.

Each participant will receive both treatments (massage gun and heat pad), but in a different order depending on group assignment. There will be a two-week washout phase between the two treatments to ensure that the effects of the first treatment do not influence the second.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate to the study
* Signed written informed consent

Exclusion Criteria:

* Inability to follow procedures or insufficient knowledge of project language, inability to give consent
* a history of drug ingestion within the past week (e.g. pain relievers, muscle relaxants, botox and anti-inflammatory drugs)
* systemic diseases
* Contraindications listed on the massage-gun instruction manual systemic and related to the use on the masseter area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Masseter muscle stiffness | The time from the first appointment to the second (final) appointment will be two weeks.
  Muscle stiffness will be assessed using shear wave elastography (SWE) via ultrasound. Results will be reported in kilopascals (kPa) and/or meters per second (m/s).

SECONDARY OUTCOMES:
Algometry of the Masseter Muscle | The time from the first appointment to the second (final) appointment will be two weeks.
  Algometry is the quantitative assessment of pain sensitivity, performed using a pressure algometer to determine pressure pain thresholds (PPTs) at specific anatomical sites.
mouth opening | The time from the first appointment to the second (final) appointment will be two weeks.
  The mouth opening will be measured with a ruler.
maximum bite force | The time from the first appointment to the second (final) appointment will be two weeks.
  Maximum bite force can be measured with a bite sensor or an occlusal force-meter, that is placed between the patients' teeth. The patient is requested to bite on the bite sensor as hard as possible. Bite force is usually measured in Newton.
chewing efficiency | The time from the first appointment to the second (final) appointment will be two weeks.
  Chewing efficiency will be measured with a two-coloured chewing gum. The person tested will take two chewing gums simultaneously, both with different colour. The gums must be chewed 20 times and after that the mass is pressed on a glass plate and is analysed how much the colours have mixed.

CONTACTS AND LOCATIONS:
Overall Officials: Mutlu Özcan, Prof. Dr. med. dent., Study Chair — University of Zurich
Locations (1):
- Zentrum für Zahnmedizin, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request from another research group, the raw IPD will be anonymized and shared.
Time Frame: starting 6 months after publication